CLINICAL TRIAL: NCT05874440
Title: Clinical Efficacy and Safety of Tenofovir Disoproxil Fumarate and Entcavir in Treatment of Chronic Hepatitis B Patients in Upper Egypt
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Rehab Abdelraof Mohamed, Clinical Efficacy and Safety of Tenofovir Disoproxil Fumarate and Entcavir in Treatment of Chronic Hepatitis B patients in Upper Egypt, Sohag University
Other Study IDs: Soh-Med-23-04-05MD
Record Dates: First submitted 2023-05-02; First posted 2023-05-24 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Chronic Hepatitis b Patients
MeSH Terms: interventions — Tenofovir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Tenofovir Disoproxil Fumarate and Entcavir — Regular registration of side effects of the drugs, cause of non-compliance to treatment

SUMMARY:
Chronic hepatitis B (CHB) is one of the major causes of chronic liver diseases worldwide. Around 296 million people were living with chronic hepatitis B infection, with 1.5 million new infections each year and more than 820 thousand people die because of hepatitis B virus (HBV) related complications

DETAILED DESCRIPTION:
Chronic Hepatitis B is a long-term liver disease. The disease is often characterized by abnormal levels of serum ALT and AST, as well as liver histology, and is transmitted through blood, sexual contact, and mother-to-child transmission.

The symptoms of CHB include fatigue, nausea, abdominal distension, and Rt hypochondrial pain, and in severe cases, it can be accompanied by chronic liver disease, spider nevus, abnormal liver function, or persistent abnormality. The progression of hepatitis B virus (HBV) is closely linked to its replication, and the most effective way to prevent it is through hepatitis B vaccination. However, there is currently no specific drug available to eliminate the virus in patients with chronic hepatitis B (CHB) due to the low rate of HBsAg clearance. Instead, primary treatment methods for CHB aim to inhibit virus replication for an extended period and delay the onset of liver cirrhosis and hepatocellular carcinoma. Antiviral, liver protection, antifibrosis, and immunomodulatory therapies are used to achieve this goal. Among these therapies, nucleoside (acid) analogs (NA) are commonly used, with drugs such as entecavir (ETV) and tenofovir (TDF) being the most effective. Tenofovir is a new type of nucleotide reverse transcriptase inhibitor, which inhibits reverse transcriptase similarly to nucleoside reverse transcriptase inhibitors. To a certain extent, it can reduce transaminase, protect the liver, and has a good effect on the treatment of hepatitis B. ETV is a carboxylic analog of 2'-deoxyguanosine, which inhibits HBV DNA polymerase by competing with natural deoxy guanosine triphosphate.

The use of entecavir (ETV) and tenofovir disoproxil (TDF) are both effective in managing hepatitis B virus (HBV) infection, and are well-tolerated by most patients.

While there are no significant differences in the ability of the various treatments to suppress the virus, some studies suggest that TDF may achieve biochemical response more quickly. Nucleoside analogs with a high barrier to resistance are unlikely to lead to the clearance of hepatitis B surface antigen, and should therefore be continued for most patients throughout their lifetime. However, there are concerns about the potential for toxicity with TDF in patients who have additional risk factors for kidney and bone problems. It is important to monitor for adverse effects, and switching to ETV may be a safe and effective alternative for patients with HBV. Although effective antiviral treatment can improve the clinical outcome of chronic HBV patients, there is still a risk of developing hepatocellular carcinoma (HCC) even with viral suppression. It is unclear whether TDF-based regimens offer any additional benefits over ETV in preventing HCC, and more research is needed in this area. Studies conducted on both TDF and ETV have demonstrated their safety in both pivotal trials and real-life cohorts. In less than 10% of cases, mild side effects such as headache, fatigue, dizziness, nausea, abdominal discomfort, and nasopharyngitis have been reported for both drugs. These side effects are generally temporary and not severe enough to require discontinuation of treatment. However, TDF has been associated with kidney dysfunction, particularly in patients with pre-existing kidney disease or other risk factors for renal impairment. Furthermore, TDF has been linked to bone disease. As a result, the European Association for the Study of the Liver recommends selecting or switching to ETV for patients with chronic hepatitis B who are at greater risk of bone and kidney toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Patient with HbsAg positivity for at least 6 months.
* Patients have HbeAg positive or negative.
* Patient recived Theryapy with ETV 0.5 or 1 mg/day or TDF 300 mg/day.
* Patients have Regular monitoring every 6 months.

Exclusion Criteria:

* Patients younger than 18 years old.
* Patients co-infected with hepatitis C, hepatitis D.
* Patients receiving immune suppressive therapy or with history of immunodeficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of individuals who have been diagnosed with CHB and have undergone treatment with either ETV or TDF. These patients will be monitored regularly to evaluate the efficacy and safety of the respective therapies. Patients who meet the inclusion criteria and do not have any of the specified exclusion criteria will be eligible to participate in the study.
  It is important to note that the study population will exclude individuals who are under 18 years old, those with co-infections of HCV or HDV, as well as patients receiving immune suppressive therapy or with a history of immunodeficiency. By defining the study population based on these criteria, the research can focus on evaluating the outcomes and safety profile of ETV and TDF in a specific group of patients with CHB.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-04-15 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Experiencing Treatment-Related Adverse Events as Assessed by CTCAE v4.0Disoproxil Fumarate and Entcavir | 12 months
  This outcome measure aims to evaluate the safety profile of Tenofovir Disoproxil Fumarate (TDF) and Entecavir (ETV) in the treatment of Chronic Hepatitis B (CHB). It will involve assessing and reporting the number of participants who experience adverse events related to the treatment, utilizing the Common Terminology Criteria for Adverse Events version 4.0 (CTCAE v4.0) for assessment
Reduction in Hepatitis B Viral Load with Entecavir (ETV) Treatment as Measured by Quantitative PCR | 12 months
  The primary outcome measure of this study is the reduction in hepatitis B viral load with Entecavir (ETV) treatment, which will be assessed using quantitative polymerase chain reaction (PCR) analysis. The viral load will be quantified by measuring the amount of hepatitis B virus DNA in the patient's blood sample. The collected measurement data will be aggregated to determine the effectiveness of Entecavir (ETV) in reducing viral replication in patients with chronic hepatitis B
Reduction in Hepatitis B Viral Load with Tenofovir Disoproxil Fumarate (TDF) Treatment as Measured by Quantitative PCR | 12 months
  The primary outcome measure of this study is the reduction in hepatitis B viral load with Tenofovir Disoproxil Fumarate (TDF) treatment, which will be assessed using quantitative polymerase chain reaction (PCR) analysis. The viral load will be quantified by measuring the amount of hepatitis B virus DNA in the patient's blood sample. The collected measurement data will be aggregated to determine the effectiveness of Tenofovir Disoproxil Fumarate (TDF) in reducing viral replication in patients with chronic hepatitis B

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University hospitals, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Choi J, Jo C, Lim YS. Tenofovir Versus Entecavir on Recurrence of Hepatitis B Virus-Related Hepatocellular Carcinoma After Surgical Resection. Hepatology. 2021 Feb;73(2):661-673. doi: 10.1002/hep.31289. Epub 2020 Nov 2. PMID 32324905
- [Background] Langley DR, Walsh AW, Baldick CJ, Eggers BJ, Rose RE, Levine SM, Kapur AJ, Colonno RJ, Tenney DJ. Inhibition of hepatitis B virus polymerase by entecavir. J Virol. 2007 Apr;81(8):3992-4001. doi: 10.1128/JVI.02395-06. Epub 2007 Jan 31. PMID 17267485
- [Background] Lim YS. Management of Antiviral Resistance in Chronic Hepatitis B. Gut Liver. 2017 Mar 15;11(2):189-195. doi: 10.5009/gnl15562. PMID 28183162
- [Background] Shi YW, Yang RX, Fan JG. Chronic hepatitis B infection with concomitant hepatic steatosis: Current evidence and opinion. World J Gastroenterol. 2021 Jul 14;27(26):3971-3983. doi: 10.3748/wjg.v27.i26.3971. PMID 34326608